CLINICAL TRIAL: NCT01124149
Title: A Phase 4, Open-label, Multicenter, Prospective Study to Evaluate the Effect of Remission Status on the Ability to Maintain or Achieve Clinical and Endoscopic Remission During a 12-Month, Long-term Maintenance Phase With 2.4g/Day MMX Mesalamine/Mesalazine Once Daily in Adult Subjects With Ulcerative Colitis
Brief Title: Ability to Maintain or Achieve Clinical and Endoscopic Remission With MMX Mesalamine Once Daily in Adults With Ulcerative Colitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPD476-409; 2009-017044-13 (EudraCT Number)
Record Dates: First submitted 2010-05-13; First posted 2010-05-14 (Estimated); Results first posted 2013-12-02 (Estimated); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Mesalamine

ARMS (1):
- MMX mesalamine/ mesalazine (Experimental)
  Interventions: Drug: MMX mesalamine/ mesalazine

INTERVENTIONS:
Drug: MMX mesalamine/ mesalazine — 4.8g/day given QD (four 1.2g tablets) for 8 weeks, 2.4g/day given QD (two 1.2g tablets) for 12 months
  Other Names: Lialda; Mezavant; Mezavant XL; Mezavant LP

SUMMARY:
This study was designed to evaluate if subjects who achieve complete remission after 8 weeks of acute therapy with MMX mesalamine/mesalazine 4.8g/day given QD have better long-term outcomes and remain in remission longer compared with subjects who demonstrate only partial remission after acute therapy with MMX mesalamine/mesalazine 4.8g/day given QD. Therefore, subjects who achieve either complete or partial remission will enter into a 12-month maintenance phase, during which they will receive MMX mesalamine/mesalazine 2.4g/day given QD. Remission status for the 2 groups will be evaluated and compared at the end of this 12-month maintenance period. The data obtained from this study will provide scientifically meaningful information to demonstrate that achieving complete remission (clinical and endoscopic remission) is important for a better long-term prognosis, or that the current paradigm of symptomatic treatment is appropriate.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged 18 or older
2. Male, or non-pregnant, non-lactating female who agrees to comply with any applicable contraceptive requirements of the protocol
3. Diagnosis of active mild to moderate UC (acute flare or newly diagnosed)
4. Stable maintenance therapy of 5-ASA less than or equal to 3.2 g/day (excluding MMX mesalamine/mesalazine), if 5-ASA is being taken at the onset of acute flare.

Exclusion Criteria:

1. Severe UC
2. Acute flare with onset greater than >6 weeks prior to baseline while on maintenance therapy. There is no limit to the onset of flare prior to baseline if the flare is untreated.
3. Acute flare while on maintenance MMX mesalamine/mesalazine (Lialda, Mezavant, Mezavant XL, Mezavant LP)
4. Unsuccessfully treated current acute flare using steroids or 5-ASA doses >3.2 g/day
5. Acute flare on a 5-ASA maintenance therapy of >3.2 g/day
6. Systemic or rectal steroids use within the 4 weeks prior to screening or immunosuppressants within the last 6 weeks prior to screening
7. History of biologic (anti-TNF agent) use
8. Antibiotic use or repeated use (>3 consecutive days of use at doses above the prescribed over-the-counter dose) of any anti-inflammatory drugs, including non-steroidal anti-inflammatory drugs such as aspirin, COX-2 inhibitors or ibuprofen, within 7 days prior to screening. However, prophylactic use of a stable dose of aspirin up to 325mg/day for cardiac disease is permitted
9. Current or recurrent disease, other than UC, that could affect the colon, the action, absorption, or disposition of the IMP, or clinical or laboratory assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 759 (Actual)
Dates: Start 2010-06-29 (Actual); Primary Completion 2012-12-07 (Actual); Study Completion 2012-12-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (105):
- United States (34):
  - Birmingham Gastroenterology Associates, PC, Birmingham, Alabama
  - Advanced Clinical Research Institute, Anaheim, California
  - Digestive & Liver Disease Specialists, Garden Grove, California
  - Long Beach VA Medical Center, Long Beach, California
  - Clinical Applications Laboratories, Inc., San Diego, California
  - Conneticut Gastroenterolgy Institute, Bristol, Connecticut
  - Borland-Groover Clinic, Jacksonville, Florida
  - United Medical Research, New Smyrna Beach, Florida
  - Advances Gastroenterology Associates, Palm Harbor, Florida
  - Atlanta Gastroenterology Associates, LLC, Atlanta, Georgia
  - Atlanta Gastroenterology Associates, Marietta, Georgia
  - University of Chicago Medical Center, Chicago, Illinois
  - Midwest Clinical Research Associates, Moline, Illinois
  - Gastrointestinal Clinic of Quad Cities, Davenport, Iowa
  - New Orleans Research Institute, Metairie, Louisiana
  - Delta Research Partners, Monroe, Louisiana
  - Louisiana Research Center, LLC, Shreveport, Louisiana
  - Digestive Disorders Associates, Annapolis, Maryland
  - Digestive Disease Associates, Baltimore, Maryland
  - Center for Digestive Health, Troy, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Center for Digestive & Liver Disease, Inc., Mexico, Missouri
  - Long Island Clinical Research Associates, LLP, Great Neck, New York
  - Gastrointestinal Research Associates, Setauket, New York
  - LeBauer Research Associates, Greensboro, North Carolina
  - Ohio Gastroenterolgy and Liver Intstitute, Cincinnati, Ohio
  - Regional Gastroenterology Associates of Lancaster, Ltd., Lancaster, Pennsylvania
  - Gastroenterology Associates, LLC, Kingsport, Tennessee
  - S.D. Khan, Houston, Texas
  - Gastroenterology Clinic of San Antonio, PA, San Antonio, Texas
  - Colon and Rectal Disease Center, Sandy City, Utah
  - Physicians Research Option, LLC, Sandy City, Utah
  - Alexandria Clinical Research, Alexandria, Virginia
  - Wisconsin Center for Advances Research, Milwaukee, Wisconsin
- Belgium (3):
  - Imelda General Hospital, Bonheiden
  - vzw AZ Groeninge, Kortrijk
  - Heilig Hart ziekenhuis vzw Roeselare-Menen, Roeselare
- Canada (5):
  - McMaster University Medical Centre, Hamilton, Ontario
  - Toronto Digestive Disease Associates, Inc., Toronto, Ontario
  - Royal Victoria Hospital, Montreal, Quebec
  - CHAUQ- Hopital du Saint-Sacrement, Québec, Quebec
  - Alpha Recherche Clinique, Québec, Quebec
- Colombia (4):
  - Hospital pablo Tobon uribe, Medellín, Antioquia
  - Promotora medica las Americas S.A., Medellín, Antioquia
  - Ugasend S.A., Barranquilla, Atlántico
  - FOQUS, Centro de Investigacion Clinica, Bogota, Cundinamarca
- Czechia (10):
  - Private Gastroenterology centre, České Budějovice
  - Derma Plus s.r.o. Gastroenterology, České Budějovice
  - Hepato-Gastroenterology HK s.r.o., Hradec Králové
  - Nemocnice Jablonec nad Nisou, Jablonec nad Nisou
  - Faculty hospital Plzen- Lochotin, Pilsen
  - IKEM (Institute klinicke a experimentalni mediciny), Prague
  - Klinicke Centrum ISCARE I.V.F., Prague
  - Nemocnice Tabor a.s., Tábor
  - Massarykova Nemocnice-Masaryk Hospital, Ústí nad Labem
  - Orlickoustecka nemocnice a.s. (Hospital), Ústí nad Orlicí
- France (3):
  - Hopital Saint Andre, Bordeaux
  - CHU Estaing, Clermont-Ferrand
  - CHU Nantes- Hotel Dieu, Nantes
- Germany (2):
  - Medizinische Hochschule Hannover/ Zentrum Innere Medizin/Gastroenterologie, Hanover
  - Stawdtisches Klinikum Lueneburg Gastroenterologie, Lüneburg
- Hungary (5):
  - Debreceni Egyetem Orvos-es Egeszsegtudomanyi Centrum III. sz. Belgyogyazati Klinika, Debrecen
  - Bekes Megyei Kepviselotestulet Pandy Kalman Korhaza, Endoszkopos laboratorium, Gyula
  - Borsod-Abauj-Zemplen Megyei Korhaz es Egyrtrmi Oktato Korhaz, II. Belgyogyaszat, Miskolc
  - Karolina Korhaz, Belgyogyaszat es Gasztroenterologia, Mosonmagyaróvár
  - Javorszky Odon Varosi Korhaz, Gasztroenterologia, Vác
- India (13):
  - Asian Institute of Gastroenterology, Hyderabad, Andhra Pradesh
  - Manikya Institute of Gastroenterology & Hepatology, Visakhapatnam, Andhra Pradesh
  - Institute of Digestive & Liver Diseases, Guwahati, Assam
  - Mehta Hospital, Ahmedabad, Gujarat
  - Kasturba Medical College Hospital, Mangalore, Kamataka
  - Sree Gokulam Medical College and Research Foundation, Thiruvananthapuram, Kerala
  - Gastroenterology & Endoscopy Centre, Nagpur, Maharashtra
  - Sahyandri Speciality Hospital, Pune, Maharashtra
  - Poona Hospital & Research Centre, Pune, Maharashtra
  - Dayanand Medical College and hospital, Ludhiana, Punjab
  - S R Kalla Memorial Gastro & General Hospital, Jaipur, Rajasthan
  - Dr. Nijhawan Clinic, Jaipur, Rajasthan
  - Chhatrapati Shahuji Maharaj Medical University, Lucknow, Uttar Pradesh
- Ireland (3):
  - Adelaide and Meath Hospital, Dublin
  - St Vincents' University Hospital, Dublin
  - Beaumont Hospital, Dublin
- Poland (7):
  - NZOZ Centrum Medyczne Szpital Sw. Rodziny, Lodz
  - NZOZ Centrum Medyczne HCP, Poznan
  - Endoskopia Sp z o.o., Sopot
  - Indyw. Spec. Prakt. Lek. w Dziedzinie Chirurgii Ogolnej i Gastroenterologii, Torun
  - Nzoz Vivamed, Warsaw
  - LexMedica, Wroclaw
  - EMC Instytut Medyczny SA, Wroclaw
- Romania (6):
  - CMI de Gastroenterologie, Târgu Mureş, Mureș County
  - Clinical Hospital "Dr. I. Cantacuzino", Bucharest
  - Institutul Clinic Fundeni, Bucharest
  - Emergency University Clinical Hospital Bucuresti, Bucharest
  - Policlinic Algomed SRL, Timișoara
  - Policlinica "Dr. Citu" SRL, Timișoara
- South Africa (7):
  - Rose Park Hospital Boanerges CC Trials, Bloemfontein, Free State
  - St. Augustine's Hospital, Durban, KwaZulu-Natal
  - Parklands Medical Centre, Durban, KwaZulu-Natal
  - Panorama Medi-Clinic, Cape Town, Western Cape
  - Louis Leipoldt Medical Centre, Cape Town, Western Cape
  - Kingsbury Hospital, Cape Town, Western Cape
  - Greenacres Hospital, Port Elizabeth
- Hospital Universitario La Princesa, Madrid, Spain
- United Kingdom (2):
  - St Mark's Hospital, Harrow, Middlesex
  - John Radcliffe Hospital, Headington, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Stevens TW, Gecse K, Turner JR, de Hertogh G, Rubin DT, D'Haens GR. Diagnostic Accuracy of Fecal Calprotectin Concentration in Evaluating Therapeutic Outcomes of Patients With Ulcerative Colitis. Clin Gastroenterol Hepatol. 2021 Nov;19(11):2333-2342. doi: 10.1016/j.cgh.2020.08.019. Epub 2020 Aug 13. PMID 32801008
- [Derived] Willian MK, D'Haens G, Yarlas A, Joshi AV. Changes in health-related quality of life and work-related outcomes for patients with mild-to-moderate ulcerative colitis receiving short-term and long-term treatment with multimatrix mesalamine: a prospective, open-label study. J Patient Rep Outcomes. 2018 Apr 27;2:22. doi: 10.1186/s41687-018-0046-5. eCollection 2018 Dec. PMID 30294708
- [Derived] Yarlas A, D'Haens G, Willian MK, Teynor M. Health-Related Quality of Life and Work-Related Outcomes for Patients With Mild-to-Moderate Ulcerative Colitis and Remission Status Following Short-Term and Long-Term Treatment With Multimatrix Mesalamine: A Prospective, Open-Label Study. Inflamm Bowel Dis. 2018 Jan 18;24(2):450-463. doi: 10.1093/ibd/izx041. PMID 29361097

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Although 639 subjects completed the Acute Phase, 167 were not eligible to enter the Maintenance Phase due to lack of efficacy and 2 others withdrew prior to entering the maintenance Phase and 1 was withdrawn per IVRS prior to entering the Mainenance Phase. Therefore, 469 subjects entered the Maintenance Phase.
Groups:
- MMX Mesalamine/ Mesalazine: 4.8g/day given QD for 8 weeks in the Acute Phase and 2.4g/day given QD for 12 months in the Maintenance Phase
Period: Acute Phase
Arm/Group | MMX Mesalamine/ Mesalazine
Started | 722
Completed | 639
Not Completed | 83
Not completed — Withdrawal by Subject | 22
Not completed — Adverse Event | 21
Not completed — Lack of Efficacy | 17
Not completed — Protocol Violation | 14
Not completed — Lost to Follow-up | 2
Not completed — Prolonged antibiotic therapy | 1
Not completed — Sponsor request | 1
Not completed — UC symptoms not ameliorated | 1
Not completed — Non-compliance | 1
Not completed — Low hemoglobin | 1
Not completed — Travelling to another country | 1
Not completed — Sponsor decision | 1
Period: Maintenance Phase
Arm/Group | MMX Mesalamine/ Mesalazine
Started | 469
Completed | 373
Not Completed | 96
Not completed — Lack of Efficacy | 40
Not completed — Adverse Event | 24
Not completed — Lost to Follow-up | 15
Not completed — Withdrawal by Subject | 10
Not completed — Protocol Violation | 5
Not completed — Coordinator error | 1
Not completed — Non-compliance | 1

BASELINE CHARACTERISTICS:
Population: The Safety Population was used. Safety Population defined as all subjects who took at least 1 dose of investigational product during the Acute or Maintenance Phase (n=717).
Arm/Group | MMX Mesalamine/ Mesalazine
Number analyzed (Participants) | 717
Age, Continuous [Mean (Standard Deviation); unit: Years] | 42.9 (13.97)
Age, Customized [Count of Participants; unit: Participants]
  >=65 years | 51
  <=18 years | 10
  Between 18 and 65 years | 656
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 308
  Male | 409
Region of Enrollment [Count of Participants; unit: Participants] — All enrolled subjects (n=722).
  Participants
    BELGIUM | 22
    CANADA | 39
    COLOMBIA | 74
    CZECH REPUBLIC | 130
    FRANCE | 2
    HUNGARY | 30
    INDIA | 200
    IRELAND | 9
    POLAND | 52
    ROMANIA | 41
    SOUTH AFRICA | 21
    SPAIN | 3
    UNITED KINGDOM | 3
    UNITED STATES | 96

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects in Complete Remission at Month 12 of Maintenance Phase
Description: Complete remission was defined as a modified Ulcerative Colitis Disease Activity Index (UC-DAI) <=1 with a score of 0 for rectal bleeding and stool frequency and at least a 1-point reduction in endoscopy score from baseline. The modified UC-DAI score is the sum of the scores of 4 parameters (stool frequency, rectal bleeding, endoscopy score, and physician global assessment), each scoring between 0 and 3, making 12 the worst score. Endoscopy score (mucosal appearance) ranges from 0-3 (0 = normal, 1 = mild , 2 = moderate, 3 = severe). Rectal bleeding is assessed on a scale from 0-3 (0 = no rectal bleeding, 1 = streaks of blood, 2 = obvious blood, 3 = mostly blood). Stool frequency is assessed on a scale of 0-2 (0 = 0-1 more than normal per day, 1 = 2-3 more than normal per day, 2 = 4 or more than normal per day).
Time Frame: 12 months
Population: Maintenance Phase Efficacy Population included all subjects who, during the Maintenance Phase, took at least 1 dose of investigational product and had at least 1 post-dose efficacy assessment.
Measure: Number; unit: percentage of subjects
Groups:
- MMX Mesalamine/ Mesalazine (Complete Remission Acute Phase): Subjects received 4.8g/day given QD for 8 weeks in the Acute Phase and were classified as having complete remission at the end of the Acute Phase. Complete (clinical and endoscopic) remission was defined as a modified UC-DAI <=1 with a score of 0 for rectal bleeding and stool frequency and at least a 1-point reduction in endoscopy score from baseline. These subjects then received 2.4g/day given QD for 12 months in the Maintenance Phase.
- MMX Mesalamine/ Mesalazine (Partial Remission Acute Phase): Subjects received 4.8g/day given QD for 8 weeks in the Acute Phase and were classified as having partial remission at the end of the Acute Phase. Partial remission was defined as a modified UC-DAI <=3 with a combined stool frequency and rectal bleeding score of <=1 and not in complete remission. These subjects then received 2.4g/day given QD for 12 months in the Maintenance Phase.
Arm/Group | MMX Mesalamine/ Mesalazine (Complete Remission Acute Phase) | MMX Mesalamine/ Mesalazine (Partial Remission Acute Phase)
Number analyzed (Participants) | 182 | 277
percentage of subjects | 47.8 | 26.0
Statistical Analysis 1: Comparison: MMX Mesalamine/ Mesalazine (Complete Remission Acute Phase) vs MMX Mesalamine/ Mesalazine (Partial Remission Acute Phase); Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.61, 95% CI 2-sided [1.76 to 3.87]

2. Secondary Outcome: Percentage of Subjects in Clinical Remission at Month 12 of Maintenance Phase
Description: Clinical remission was defined as a score of 0 for rectal bleeding and stool frequency. Rectal bleeding is assessed on a scale from 0-3 (0 = no rectal bleeding, 1 = streaks of blood, 2 = obvious blood, 3 = mostly blood). Stool frequency is assessed on a scale of 0-2 (0 = 0-1 more than normal per day, 1 = 2-3 more than normal per day, 2 = 4 or more than normal per day).
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | MMX Mesalamine/ Mesalazine (Complete Remission Acute Phase) | MMX Mesalamine/ Mesalazine (Partial Remission Acute Phase)
Number analyzed (Participants) | 182 | 277
percentage of subjects | 58.8 | 40.4
Statistical Analysis 1: Comparison: MMX Mesalamine/ Mesalazine (Complete Remission Acute Phase) vs MMX Mesalamine/ Mesalazine (Partial Remission Acute Phase); Test type: Superiority or Other; p < 0.001, Regression, Logistic; Odds Ratio (OR) = 2.10, 95% CI 2-sided [1.44 to 3.07]

3. Secondary Outcome: Relapse in Ulcerative Colitis at Month 12 of Maintenance Phase
Description: Relapse was defined in the Maintenance Phase as the need for alternative treatment for UC (including surgery); subjects were classified as having a relapse if they had withdrawn from the study due to a lack of efficacy.
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | MMX Mesalamine/ Mesalazine (Complete Remission Acute Phase) | MMX Mesalamine/ Mesalazine (Partial Remission Acute Phase)
Number analyzed (Participants) | 182 | 277
percentage of subjects | 6.0 | 10.5

4. Secondary Outcome: Percentage of Subjects With Mucosal Healing at 12 Months of Maintenance Phase
Description: Subjects with mucosal healing were defined as subjects who had an endoscopy score <=1. Endoscopy score (mucosal appearance) ranges from 0-3 (0 = normal, 1 = mild , 2 = moderate, 3 = severe).
Time Frame: 12 months
Population: as for outcome 1
Measure: Number; unit: percentage of subjects
Arm/Group | MMX Mesalamine/ Mesalazine (Complete Remission Acute Phase) | MMX Mesalamine/ Mesalazine (Partial Remission Acute Phase)
Number analyzed (Participants) | 182 | 277
percentage of subjects | 76.4 | 63.5

5. Secondary Outcome: Improvement in Rectal Bleeding Score During the Acute Phase
Description: Improvement was defined as at least a 1-point reduction in the rectal bleeding score from baseline at each assessment point. Rectal bleeding is assessed on a scale from 0-3 (0 = no rectal bleeding, 1 = streaks of blood, 2 = obvious blood, 3 = mostly blood).
Time Frame: 3 and 8 weeks
Population: Acute Phase Safety Population included all subjects who, during the Acute Phase, took at least 1 dose of investigational product.
Measure: Number; unit: percentage of subjects
Groups:
- MMX Mesalamine/ Mesalazine: 4.8g/day given QD for 8 weeks in the Acute Phase
Arm/Group | MMX Mesalamine/ Mesalazine
Number analyzed (Participants) | 717
percentage of subjects
  Week 3 | 42.4
  Week 8 | 59.8

6. Secondary Outcome: Improvement in Stool Frequency Symptoms During the Acute Phase
Description: Improvement was defined as at least a 1-point reduction in the stool frequency score from baseline at each assessment point. Stool frequency is assessed on a scale of 0-2 (0 = 0-1 more than normal per day, 1 = 2-3 more than normal per day, 2 = 4 or more than normal per day).
Time Frame: 3 and 8 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | MMX Mesalamine/ Mesalazine
Number analyzed (Participants) | 717
percentage of subjects
  3 Weeks | 38.5
  8 Weeks | 58.9

7. Secondary Outcome: Percentage of Subjects in Complete Remission at Week 8 of Acute Phase
Description: Complete (clinical and endoscopic) remission was defined as a modified UC-DAI <=1 with a score of 0 for rectal bleeding and stool frequency and at least a 1-point reduction in endoscopy score from baseline. The modified UC-DAI score is the sum of the scores of 4 parameters (stool frequency, rectal bleeding, endoscopy score, and physician global assessment), each scoring between 0 and 3, making 12 the worst score. Endoscopy score (mucosal appearance) ranges from 0-3 (0 = normal, 1 = mild , 2 = moderate, 3 = severe). Rectal bleeding is assessed on a scale from 0-3 (0 = no rectal bleeding, 1 = streaks of blood, 2 = obvious blood, 3 = mostly blood). Stool frequency is assessed on a scale of 0-2 (0 = 0-1 more than normal per day, 1 = 2-3 more than normal per day, 2 = 4 or more than normal per day).
Time Frame: 8 Weeks
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | MMX Mesalamine/ Mesalazine
Number analyzed (Participants) | 717
percentage of subjects | 25.9

8. Secondary Outcome: Percentage of Subjects in Partial Remission at Week 8 of Acute Phase
Description: Partial remission was defined as a modified UC-DAI <=3 with a combined stool frequency and rectal bleeding score of <=1 and not in complete remission. The modified UC-DAI score is the sum of the scores of 4 parameters (stool frequency, rectal bleeding, endoscopy score, and physician global assessment), each scoring between 0 and 3, making 12 the worst score. Endoscopy score (mucosal appearance) ranges from 0-3 (0 = normal, 1 = mild , 2 = moderate, 3 = severe). Rectal bleeding is assessed on a scale from 0-3 (0 = no rectal bleeding, 1 = streaks of blood, 2 = obvious blood, 3 = mostly blood). Stool frequency is assessed on a scale of 0-2 (0 = 0-1 more than normal per day, 1 = 2-3 more than normal per day, 2 = 4 or more than normal per day).
Time Frame: 8 weeks
Population: as for outcome 5
Measure: Number; unit: percentage of subjects
Arm/Group | MMX Mesalamine/ Mesalazine
Number analyzed (Participants) | 717
percentage of subjects | 39.3

ADVERSE EVENTS:
Groups:
- MMX Mesalamine/ Mesalazine (Acute Phase): 4.8g/day given QD for 8 weeks in the Acute Phase
- MMX Mesalamine/ Mesalazine (Maintenance Phase): 2.4 g/day given QD for 12 months in the Maintenance Phase
Arm/Group | MMX Mesalamine/ Mesalazine (Acute Phase) | MMX Mesalamine/ Mesalazine (Maintenance Phase)
Serious Adverse Events (participants affected / at risk) | 13/717 | 14/461
Other Adverse Events (participants affected / at risk) | 60/717 | 65/461
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MMX Mesalamine/ Mesalazine (Acute Phase) (N=717) | MMX Mesalamine/ Mesalazine (Maintenance Phase) (N=461)
Myocardial infarction (Cardiac disorders) | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 2 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Arthritis bacterial (Infections and infestations) | 1 | 0
Lung infection (Infections and infestations) | 1 | 0
Pneumonia staphylococcal (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 0
HIV test positive (Investigations) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 1
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 1 | 0
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 0 | 2
Atrial fibrillation (Cardiac disorders) | 0 | 1
Bundle branch block left (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Diarrhea (Gastrointestinal disorders) | 0 | 3
Pyrexia (General disorders) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 2
C-reactive protein increased (Investigations) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Hemorrhagic stroke (Nervous system disorders) | 0 | 1
Radiculopathy (Nervous system disorders) | 0 | 1
Metrorrhagia (Reproductive system and breast disorders) | 0 | 1
Venous thrombosis limb (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MMX Mesalamine/ Mesalazine (Acute Phase) (N=717) | MMX Mesalamine/ Mesalazine (Maintenance Phase) (N=461)
Colitis ulcerative (Gastrointestinal disorders) | 10 | 43
Drug ineffective (General disorders) | 50 | 22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If a multicenter publication is not submitted within twelve (12) months after conclusion, abandonment or termination of the Study at all sites, or after Sponsor confirms there shall be no multicenter Study publication, the Institution and/or such Principal Investigator may publish the results from the Institution site individually.